CLINICAL TRIAL: NCT05931887
Title: Evaluation of the Novel Silq ClearTract Catheter in Patients With Chronic Urinary Retention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Silq Technologies Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: STC002
Record Dates: First submitted 2023-06-16; First posted 2023-07-05 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Catheter Infection; Catheter Blockage; Catheter Related Complication; Catheter Calcification

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- SILQ ClearTract 100% Silicone 2-Way Foley Catheter (Active Comparator): Subjects in this arm will receive the SILQ ClearTract 100% Silicone 2-Way Foley Catheter for approximately the first 3 month period of enrollment. In a subsequent period of approximately 3 months subjects in this arm will receive their current standard of care catheter.
  Interventions: Device: SILQ ClearTract 100% Silicone 2-Way Foley Catheter
- Standard of Care Catheter (Active Comparator): Subjects in this arm will receive their current Standard of Care Catheter for the first 3 month period of enrollment. In a subsequent period of approximately 3 months subjects in this arm will receive the SILQ ClearTract 100% Silicone 2-Way Foley Catheter
  Interventions: Device: SILQ ClearTract 100% Silicone 2-Way Foley Catheter

INTERVENTIONS:
Device: SILQ ClearTract 100% Silicone 2-Way Foley Catheter — A foley catheter is assigned and used according to regular standard of care

SUMMARY:
To assess the ability of the Silq ClearTract™ 100% Silicone 2-Way Foley Catheter to reduce catheter associated complications in subjects that require a long-term indwelling Foley catheter when compared to other commercially available Foley catheters.

DETAILED DESCRIPTION:
A prospective, randomized, multi-center, post-market study in subjects that require a long-term indwelling Foley catheter.

Neurogenic bladder is commonly managed with indwelling catheters (urethral or suprapubic). Indwelling catheters are associated with multiple complications, including recurrent urinary tract infections and catheter obstruction. A randomly assigned catheter will be inserted using standard techniques. The assigned catheters will either be the SILQ ClearTract 100% Silicone 2-Way Foley Catheter or the current standard of care catheter. Subjects will continue to use the assigned catheter for a period of approximately 3 months following regular standard of care. Subjects will then be assigned the alternative catheter for an additional 3 month period after which they will be exited from the study

The purpose of the study is to compare the incidence of catheter-related complications between the SILQ treated catheter and the current standard of care catheter(s). Because these complications lead to more frequent interventions and associated treatment costs, the study will also calculate the economic impact of the use of SILQ treated catheters compared to standard of care catheters. Patient-reported outcomes will also be measured via questionnaires upon each study visit. Explanted catheter samples will also be sent to a core lab for quantification of the calcification present on the catheter surface.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Requirement of a 14 Fr, 16Fr, or 18Fr indwelling urethral or suprapubic urinary catheter (for at least 6 months) for bladder drainage.
* Able and willing to comply with study procedures
* Able and willing to give informed consent.

Exclusion Criteria:

* History of reconstructive bladder surgery such as bladder augmentation or continent catheterizable stoma.
* Cognitive deficit limiting the ability to respond to clinical questionnaires.
* Allergy or sensitivity to any catheter material used in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-07-26 (Actual); Primary Completion 2025-05-26 (Estimated); Study Completion 2025-07-26 (Estimated)

PRIMARY OUTCOMES:
Number of Catheter Related Complications | 6 months
  Catheter Related Complications can be classified as:
  i. Symptomatic Catheter Associated Urinary Tract Infection ii. Catheter Blockage iii. General Premature Interventions: Patient sought care for a catheter-related issue prior to their scheduled catheter exchange

SECONDARY OUTCOMES:
Catheter Related Complication Treatment Costs | 6 months
  All data related to complications and associated treatments will be tabulated. Corresponding treatment costs for each complication will be tabulated.
Catheter Encrustation | 6 months
  Quantitative chemical and gravimetric analysis of encrustation of removed catheters
Patient Preference | 4 months
  During the first exchange after the crossover, subjects will be asked which catheter they would prefer to continue to use
Patient Satisfaction | 6 months
  Pain and discomfort will be assessed upon each foley catheter removal using a 5 point scale. A score of 1 indicates no pain or discomfort and a score of 5 indicates severe pain or discomfort.

CONTACTS AND LOCATIONS:
Overall Officials: Evgeniy Kreydin, M.D., Principal Investigator — Rancho Los Amigos National Rehabilitation Center
Locations (1):
- Rancho Los Amigos National Rehabilitation Center, Downey, California, United States

IPD SHARING:
Plan to Share IPD: No